CLINICAL TRIAL: NCT04128904
Title: In Vitro Fertilisation Versus Intracytoplasmic Sperm Injection in Patients Without Severe Male Factor Infertility (INVICSI): a Randomised, Controlled, Multicentre Trial
Brief Title: In Vitro Fertilisation Versus Intracytoplasmic Sperm Injection in Patients Without Severe Male Factor Infertility
Acronym: INVICSI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Copenhagen University Hospital, Hvidovre (Other)
Responsible Party: Principal Investigator, Nina la Cour Freiesleben, Chief Consultant, Ph.D., Clinical Associate Professor, Copenhagen University Hospital, Hvidovre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INVICSI2019
Record Dates: First submitted 2019-10-07; First posted 2019-10-16 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2024-02

CONDITIONS: Infertility
Keywords: Infertility; Non-male factor infertility; In vitro fertilisation (IVF); Intracytoplasmic sperm injection (ICSI); Assisted reproductive technologies (ART); Live birth rate; Reproductive outcome
MeSH Terms: conditions — Infertility | interventions — Sperm Injections, Intracytoplasmic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard in vitro fertilisation (IVF) (Active Comparator): Oocytes are fertilised with standard IVF. For details please see "Project Description".
  Interventions: Procedure: IVF
- Intracytoplasmic sperm injection (ICSI) (Active Comparator): Oocytes are fertilised with ICSI. For details please see "Project Description".
  Interventions: Procedure: ICSI

INTERVENTIONS:
Procedure: IVF — Fertilisation with standard in vitro fertilisation (IVF). For details please see "Project Description".
  Arms: Standard in vitro fertilisation (IVF)
Procedure: ICSI — Fertilisation with intracytoplasmic sperm injection (ICSI). For details please see "Project Description".
  Arms: Intracytoplasmic sperm injection (ICSI)

SUMMARY:
Over recent decades, the use of intracytoplasmic sperm injection (ICSI) has increased, even among patients without severe male factor infertility. Despite the increasing use, there is no evidence to support that ICSI results in a higher live birth rate compared to conventional in vitro fertilisation (IVF) in cases without severe male factor infertility. The primary objective of this trial is to determine whether ICSI is superior to standard IVF in patients without severe male factor infertility. The primary outcome measure is live birth rate.

A total of 824 participants with infertility without severe male factor will be included in the study and allocated randomly into two groups (IVF or ICSI). The main inclusion criteria for the women are age 18-42 years, normal to slightly decreased male partner sperm/ use of donor sperm and no prior fertility treatment. In addition to live birth rate, outcome measures include fertilisation rate, total fertilisation failure, embryo quality, clinical pregnancy, miscarriage rate, preterm delivery, birth weight and congenital anomalies of the child.

The study will be performed in accordance with the ethical principles in the Helsinki Declaration. The study is approved by the Scientific Ethical Committee of the Capital Region of Denmark and the Knowledge Centre on Data Protection Compliance. Study findings will be presented in international conferences and submitted for publication in peer-reviewed journals.

DETAILED DESCRIPTION:
Background

All over the world the use of intracytoplasmic sperm injection (ICSI) with the injection of a single spermatozoon into an oocyte has gradually increased since the first report of an ICSI conceived child more than 25 years ago (Palermo et al. 1992). The latest reports from the European Society of Human Reproduction and Embryology (ESHRE) and The International Committee Monitoring Assisted Reproductive Technologies (ICMART) show that standard IVF is now used in one-third of fresh assisted reproductive technology (ART) cycles, whereas ICSI accounts for as much as two-thirds of the cycles (Dyer et al. 2016, Calhaz-Jorge et al. 2017). ICSI was initially used in fertility treatment with severe male factor infertility. However, over the years a shift towards using ICSI for other indications such as unexplained infertility, mixed factor infertility or mild male factor infertility has happened (Boulet et al., 2015; Dyer et al., 2016). Today, there is no clear evidence that using ICSI over conventional IVF in cases with non-male factor infertility yields better results (van Rumste et al., 2003). In a randomised controlled trial (RCT) from 2001 including 415 couples, better fertilisation and implantation rates after conventional IVF compared to ICSI was reported (Bhattacharya et al., 2001). In contrast, another earlier prospective study including 35 women age 21-44 years, found a better fertilisation rate after ICSI compared to sibling oocytes treated with standard IVF (Khamsi et al., 2001). A retrospective study including 745 women with non-male factor infertility reported no advantage of ICSI over conventional IVF in women aged 40 years or older (Tannus et al., 2017). In line with this, so-called poor responders with a single oocyte retrieved was shown to have similar reproductive outcomes after IVF and ICSI in a retrospective study from 2015 (Sfontouris et al., 2015). RCTs comparing outcomes after IVF and ICSI in couples/women in fertility treatment with other indications than severe male factor infertility and with live birth rate as the primary endpoint are entirely missing. Despite this, the use of ICSI in this population continuous to increase.

Therefore, a carefully designed RCT to determine whether ICSI results in higher live birth rates compared with standard IVF in patients without severe male factor infertility is warranted.

Methods

Study design:

This study is a multicentre, randomised, controlled trial with six public fertility clinics in Denmark participating. All clinics are part of a university hospital setting and all hospitals perform standardised treatments according to the public health care system in Denmark.

Participants:

All women referred for their first fertility treatment at four public fertility clinics in Denmark will be screened for eligibility. Please see criteria for eligible patients under "Eligibility".

Screening and inclusion:

Patients who are potentially eligible will receive verbal and written information about the study by the investigators during their first consultation in the fertility clinic. Inclusion and randomisation of participants to either ICSI or conventional IVF will take place after the ovulation trigger has been prescribed and before the IVF/ICSI procedure. Women/couples who wish to participate in the trial are asked to sign an informed consent form prior to enrolment. They will have a minimum of two days between receiving the information and deciding whether they wish to participate in the study or not.

Randomisation and data management:

An independent statistician has prepared a computer-generated randomisation scheme in a I:I ratio between the two arms (IVF and ICSI) ensuring concealment of treatment allocation. Permuted blocks of variable size between 4 and 12 are used for randomisation. The randomisation scheme is stratified by fertility clinic and age (three age groups: 18-25, 26-37 and 38-41) to ensure that the number of participants receiving IVF and ICSI is closely balanced within each stratum.

A designated physician or nurse from each study site is appointed. The appointed nurse/physician obtains the allocation of new patients being enrolled on their trial site. The allocation is obtained in the online platform REDCap which is also used for data collection during the study. The REDCap database has a complete audit trail and is based on anonymous subject ID numbers used in the trial.

Statistical analysis:

ITT analysis and per-protocol analysis will be performed. Baseline characteristics and outcomes will be compared using t-test, Mann-Whitney U test or chi-square tests for continuous and categorical variables or logistic regression analysis, controlling for possible confounding effects where appropriate. P-values of ≤ 0.05 will be considered statistically significant. Statistical analyses will be performed by an investigator together with statistical experts. The primary RCT analysis will be performed by an independent statistician blinded to group allocation.

Sample size calculation:

The rate of first live births after transfer of up to all of the transferable embryos from the first OPU is set to 45% in the conventional IVF group and 55 % in the ICSI group. This is a superiority trial with a power of 80% and a 2-sided p-value of 5%. The sample size is estimated to be 392 patients in each group. Post-randomization exclusion is expected to be 5%, resulting in a total of 824 patients.

Intervention:

The participants will receive conventional IVF or ICSI treatment as determined by randomisation. Both treatments are part of standard treatment regimens at the trial sites.

The fertility treatment:

The women have been treated in either a short gonadotropin-releasing hormone (GnRH)-antagonist protocol or a long GnRH-agonist protocol for ovarian stimulation. Both the controlled ovarian stimulation, transvaginal ultrasound examinations and the ovulation triggering are done according to the usual daily practice at the trial sites with ovulation trigger prescribed when a minimum of two to three follicles measure 17 mm or more. Women with only one mature follicle may also be prescribed the ovulation trigger.

OPU is performed 36±2 hours after the ovulation trigger is administered. Oocyte insemination will be IVF or ICSI according to randomisation, using established procedures at the trial sites. However, short time insemination in the IVF arm is not allowed. Embryo culture and luteal phase support will follow the usual procedures at each trial site. Blastocyst transfer is performed on day 5. Patients with a poor ovarian reserve and few oocytes retrieved (≤4) are allowed transfer day 2 or 3 according to clinical practice. Single embryo transfers are planned. Surplus blastocysts of good quality are vitrified on day 5 or 6. Transfer and cryopreservation are done according to usual practice at each trial site. In cases with total freeze of all blastocysts due to the risk of ovarian hyperstimulation syndrome (OHSS), women are not excluded from the trial. In cases where all blastocysts or spare blastocysts are vitrified these are transferred in subsequent FET cycles according to the daily practice at each trial site (i.e., natural cycles, substituted or stimulated FET cycles).

Urine pregnancy test or a serum pregnancy test is done 11-16 days after embryo transfer. If pregnancy is achieved, a transvaginal ultrasound scan is performed at pregnancy week 7-9 to confirm an ongoing and intrauterine pregnancy.

Women will be asked to inform the clinic of the result of the pregnancy as is the usual procedure in the clinic.

Outcomes:

Please see "Outcome measures".

Side effects / risks:

Both IVF and ICSI are routinely used in the clinic for fertilising the oocytes. The risk of poor or no fertilisation of the oocytes exists for both IVF and ICSI. Since both fertilisation methods are a part of standard treatment in the fertility clinics, the risk for study participants is not considered higher compared with patients who do not participate in the study.

Ethics and approvals:

The study will be performed in accordance with the ethical principles in the Helsinki Declaration.

For approvals please see "Oversight".

ELIGIBILITY:
Inclusion Criteria:

* Women 18-42 years of age (both included) at the beginning of the ovarian stimulation
* BMI 18-35 kg/m2
* Indication for IVF due to tubal factor infertility, unexplained infertility, PCOS or light to moderate decreased semen quality
* Women treated with gonadotrophin in a standard short or long protocol and receiving ovulation trigger for oocyte pick up
* First treatment cycle for the couple
* Male partner with normal or non-severely decreased sperm parameters, where the sperm sample (purified) on the day of oocyte pick up is expected to contain a minimum of 2 million/mL progressive motile spermatozoa. Alternatively use of donorsperm.
* Willing to sign the informed consent

Exclusion Criteria:

* Ovarian cysts >4 cm
* Known liver or kidney disease
* Previous IVF or ICSI treatment with current partner
* Use of donor oocytes or frozen oocytes
* Unregulated thyroid disease
* Endometriosis stage 3-4
* Hypogonadotropic hypogonadism
* Severe comorbidity (e.g. diabetes or cardiovascular disease)
* Not speaking / understanding Danish or English language
* Not willing to sign the informed consent

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 824 (Estimated)
Dates: Start 2019-11-29 (Actual); Primary Completion 2023-12-14 (Actual); Study Completion 2027-12-14 (Estimated)

PRIMARY OUTCOMES:
Cumulative live birth rate from first live birth episode of a study cycle | Minimum follow-up time is one year after inclusion
  The cumulative first live birth from the oocyte collection. Includes transfer of fresh embryos and frozen-thawed embryos.

SECONDARY OUTCOMES:
Fertilisation rate | 16-20 hours after IVF/ICSI
  Fertilisation rate per aspirated oocyte retrieved. Defined as the appearance of 2 pronuclei (PN)
Total fertilisation failure | 16-20 hours after IVF/ICSI
  Cycles with total fertilisation failure
Embryo quality | Up to six days after oocyte pick-up
  Good quality blastocysts according to Gardner classification
Time-lapse kinetics | Minimum follow-up time is one year after inclusion
  Embryo time-lapse kinetics including cleavage patterns
Embryo utilisation rate | Up to six days after oocyte pick-up
  Number of transferred + cryopreserved embryos per number of 2 PN zygotes
Cryopreservation | Up to six days after oocyte pick-up
  Number of cryopreserved blastocysts
Positive pregnancy test | 11-21 days after embryo transfer
  Positive urine or serum hCG
Multiple pregnancy | Up to 12 weeks after embryo transfer
  Number of intrauterine gestations
Ongoing pregnancy per transfer | In gestational week 7-8
  Fetal heartbeat on ultrasound
Cumulative pregnancy rates | Minimum follow-up time is one year after inclusion
  The totality of clinical pregnancies following successive treatments. This includes transfer of fresh embryos and up to all cryopreserved-thawed embryos from the first stimulation cycle if pregnancy is not achieved by the initial fresh transfer.
Biochemical pregnancy | 11-21 days after embryo transfer
  Positive urine or serum hCG without any clinical signs of intra- or extrauterine pregnancy
Pregnancy loss rate | Minimum follow-up time is one year after inclusion
  Spontaneous or planned abortions
PUL | Minimum follow-up time is one year after inclusion
  Pregnancy of unknown location
Ectopic pregnancy | Minimum follow-up time is one year after inclusion
  Pregnancy outside the uterus
Preterm delivery | Minimum follow-up time is one year after inclusion
  Delivery before gestational week 37.
Birth weight /weight for gestational age. | Minimum follow-up time is one year after inclusion
  Weight of the baby
Congenital anomaly | Minimum follow-up time is one year after inclusion
  Diagnosed congenital anomalies. Diagnosed at birth.
All live birth episodes | Minimum follow-up time is one year after inclusion
  All live births from the study oocyte collection including second and further live births
Biochemical pregnancy | Minimum follow-up time is one year after inclusion
  Positive urine or serum hCG 11-21 days after embryo transfer without any clinical signs of intra- or extrauterine pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Nina la Cour Freiesleben, ph.d., Principal Investigator — The Fertility Clinic, Hvidovre Hospital, Copenhagen University Hospital
Locations (6):
- Denmark (6):
  - The Fertility Clinic, Rigshospitalet, Copenhagen University Hospital, Copenhagen
  - The Fertility Clinic, Herlev Hospital, Copenhagen University Hospital, Herlev
  - The Fertility Clinic, Nordsjællands Hospital, Hillerød, Hillerød
  - The Fertility Clinic, the Reginal Hospital Horsens, Horsens
  - The Fertility Clinic, Hvidovre Hospital, Copenhagen University Hospital, Hvidovre
  - The Fertility Clinic, Zealand University Hospital, Køge

IPD SHARING:
Plan to Share IPD: Yes
All the individual participant data collected during the trial will be shared after deidentification upon request.
  Study protocol, Statistical analysis plan, informed consent forms, clinical study report and analytic code will be available upon request.
  Data will be available from 3 months following first publication and ending 5 years after the study has been concluded.
  Individual participant data will be shared with researches who provide a methodologically sound proposal and whose proposed use of the data has been approved by an independent review committee.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available from 3 months following first publication and ending 5 years after the study has been concluded.
Access Criteria: Individual participant data will be shared with researches who provide a methodologically sound proposal and whose proposed use of the data has been approved by an independent review committee.

REFERENCES:
- [Background] Palermo G, Joris H, Devroey P, Van Steirteghem AC. Pregnancies after intracytoplasmic injection of single spermatozoon into an oocyte. Lancet. 1992 Jul 4;340(8810):17-8. doi: 10.1016/0140-6736(92)92425-f. PMID 1351601
- [Background] Dyer S, Chambers GM, de Mouzon J, Nygren KG, Zegers-Hochschild F, Mansour R, Ishihara O, Banker M, Adamson GD. International Committee for Monitoring Assisted Reproductive Technologies world report: Assisted Reproductive Technology 2008, 2009 and 2010. Hum Reprod. 2016 Jul;31(7):1588-609. doi: 10.1093/humrep/dew082. Epub 2016 May 20. PMID 27207175
- [Background] European IVF-monitoring Consortium (EIM); European Society of Human Reproduction and Embryology (ESHRE); Calhaz-Jorge C, De Geyter C, Kupka MS, de Mouzon J, Erb K, Mocanu E, Motrenko T, Scaravelli G, Wyns C, Goossens V. Assisted reproductive technology in Europe, 2013: results generated from European registers by ESHRE. Hum Reprod. 2017 Oct 1;32(10):1957-1973. doi: 10.1093/humrep/dex264. PMID 29117383
- [Background] Boulet SL, Mehta A, Kissin DM, Warner L, Kawwass JF, Jamieson DJ. Trends in use of and reproductive outcomes associated with intracytoplasmic sperm injection. JAMA. 2015 Jan 20;313(3):255-63. doi: 10.1001/jama.2014.17985. PMID 25602996
- [Background] van Rumste MM, Evers JL, Farquhar CM. Intra-cytoplasmic sperm injection versus conventional techniques for oocyte insemination during in vitro fertilisation in patients with non-male subfertility. Cochrane Database Syst Rev. 2003;(2):CD001301. doi: 10.1002/14651858.CD001301. PMID 12804403
- [Background] Bhattacharya S, Hamilton MP, Shaaban M, Khalaf Y, Seddler M, Ghobara T, Braude P, Kennedy R, Rutherford A, Hartshorne G, Templeton A. Conventional in-vitro fertilisation versus intracytoplasmic sperm injection for the treatment of non-male-factor infertility: a randomised controlled trial. Lancet. 2001 Jun 30;357(9274):2075-9. doi: 10.1016/s0140-6736(00)05179-5. PMID 11445099
- [Background] Khamsi F, Yavas Y, Roberge S, Wong JC, Lacanna IC, Endman M. Intracytoplasmic sperm injection increased fertilization and good-quality embryo formation in patients with non-male factor indications for in vitro fertilization: a prospective randomized study. Fertil Steril. 2001 Feb;75(2):342-7. doi: 10.1016/s0015-0282(00)01674-5. PMID 11172837
- [Background] Tannus S, Son WY, Gilman A, Younes G, Shavit T, Dahan MH. The role of intracytoplasmic sperm injection in non-male factor infertility in advanced maternal age. Hum Reprod. 2017 Jan;32(1):119-124. doi: 10.1093/humrep/dew298. Epub 2016 Nov 16. PMID 27852688
- [Background] Sfontouris IA, Kolibianakis EM, Lainas GT, Navaratnarajah R, Tarlatzis BC, Lainas TG. Live birth rates using conventional in vitro fertilization compared to intracytoplasmic sperm injection in Bologna poor responders with a single oocyte retrieved. J Assist Reprod Genet. 2015 May;32(5):691-7. doi: 10.1007/s10815-015-0459-5. Epub 2015 Mar 11. PMID 25758990
- [Derived] Berntsen S, Zedeler A, Grondahl ML, Gabrielsen AV, Petersen MR, Skipper DF, Nohr B, Englund AL, Lokkegaard E, Praetorius L, Westergaard D, Pinborg A, Nielsen HS, la Cour Freiesleben N. Early embryo developmental kinetics following IVF versus ICSI in patients without severe male factor infertility: a secondary analysis of a multicentre, randomized controlled trial (INVICSI). Hum Reprod. 2025 Oct 1;40(10):1877-1885. doi: 10.1093/humrep/deaf157. PMID 40796141
- [Derived] Berntsen S, Zedeler A, Nohr B, Ronn Petersen M, Grondahl ML, Andersen LF, Lossl K, Lokkegaard E, Englund AL, Vestergaard Gabrielsen A, Praetorius L, Behrendt-Moller I, Langhoff Thuesen L, Vomstein K, Petri Lauritsen M, Ivanoska Trajcevski A, Froding Skipper D, Westergaard D, Pinborg A, Svarre Nielsen H, la Cour Freiesleben N. IVF versus ICSI in patients without severe male factor infertility: a randomized clinical trial. Nat Med. 2025 Jun;31(6):1939-1948. doi: 10.1038/s41591-025-03621-x. Epub 2025 Apr 11. PMID 40217077
- [Derived] Berntsen S, Nohr B, Grondahl ML, Petersen MR, Andersen LF, Englund AL, Knudsen UB, Praetorius L, Zedeler A, Nielsen HS, Pinborg A, Freiesleben NC. In vitro fertilisation (IVF) versus intracytoplasmic sperm injection (ICSI) in patients without severe male factor infertility: study protocol for the randomised, controlled, multicentre trial INVICSI. BMJ Open. 2021 Jun 24;11(6):e051058. doi: 10.1136/bmjopen-2021-051058. PMID 34168037